CLINICAL TRIAL: NCT02293213
Title: Utilizing Electronic Medical Record Referrals for Teratogen and Contraceptive Counseling for Women Taking Category D or X Medications: A Randomized Controlled Trial
Brief Title: EMR Referrals for Teratogen and Contraceptive Counseling for Category D or X Medication Users: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Faculty, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 130695
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Chemical Teratogen Exposure; Contraception Behavior; Contraception
Keywords: Category D; Category X; Electronic Medical Records; Long Acting Reversible Contraception
MeSH Terms: conditions — Contraception Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling only (Active Comparator): All participants who receive EMR referral to CTIS because they are taking class D or X medications AND are randomized to counseling only will receive: CTIS Counseling, Baseline Questionnaire, 3 Month Follow up Questionnaire, and 6 Month Follow up Questionnaire.
  Interventions: Behavioral: EMR Referral; Behavioral: CTIS Counseling; Behavioral: Baseline Questionnaire; Behavioral: 3 Month Follow Up Questionnaire; Behavioral: 6 Month Follow Up Questionnaire
- Counseling + Contraception Appointment (Experimental): All participants who receive EMR referral to CTIS because they are taking class D or X medications AND are randomized to counseling + Contraception Appointment will receive: CTIS Counseling, Baseline Questionnaire, Contraception Provision Appointment, 3 Month Follow up Questionnaire, and 6 Month Follow up Questionnaire.
  Interventions: Behavioral: EMR Referral; Behavioral: CTIS Counseling; Behavioral: Baseline Questionnaire; Behavioral: Contraception Provision Appointment; Behavioral: 3 Month Follow Up Questionnaire; Behavioral: 6 Month Follow Up Questionnaire

INTERVENTIONS:
Behavioral: EMR Referral — EMR referral to California Teratogen Information Services (CTIS) for use of category D or X medication.
Behavioral: CTIS Counseling — Counseling from MotherToBaby teratogen information specialist.
Behavioral: Baseline Questionnaire — Baseline Questionnaire capturing contraceptive use immediately after counseling with MotherToBaby
Behavioral: Contraception Provision Appointment — Appointment with contraception provider to discuss contraception options.
  Arms: Counseling + Contraception Appointment
Behavioral: 3 Month Follow Up Questionnaire — Questionnaire 3 months after CTIS counseling to assess contraception use and plans
Behavioral: 6 Month Follow Up Questionnaire — Questionnaire 6 months after CTIS counseling to assess contraception use and plans

SUMMARY:
Investigators propose a randomized controlled trial of women taking category D or X medications seen in family medicine, internal medicine or in the Coumadin Clinic. Women in the intervention group will receive an electronic medical record referral for teratogen counseling and contraceptive counseling with a follow up contraceptive provision appointment. The contraceptive counseling will be adapted from The Contraceptive CHOICE Project script and promote the use of the long acting reversible contraception. The women in the control group will also receive an electronic medical record referral and receive the teratogen counseling but only be told that it is important to avoid becoming pregnant. An initial survey will assess contraceptive knowledge and utilization. In addition, there will be telephone survey at 3 months and 6 months to assess contraceptive utilization and continuation.

DETAILED DESCRIPTION:
Approximately 6% of pregnancies in the United States are exposed to potentially teratogenic medications. Birth defects due to prenatal exposure to teratogenic medications are among the only truly preventable types of congenital anomalies. However, despite the risk of unintended pregnancies exposed to potentially teratogenic medications, women prescribed category D or X medications do not use more effective contraception then the general population. These women also are not more compliant with short acting methods such as oral contraceptives. The electronic medical record provides an unique opportunity to identify women taking potentially teratogenic medications and offer interdisciplinary teratogen and contraceptive counseling. These women specifically may benefit from more counseling about long acting reversible contraception while they are taking a potentially teratogenic medication.

Previous studies have revealed that women want more counseling regarding a potentially teratogenic medication when it is prescribed even if they are not planning a pregnancy or sexually active. In addition to desiring more teratogen counseling, these women may benefit from more contraceptive counseling. Eisenberg et al. identified that time constraint is one of the major barriers to providing adequate contraceptive counseling by an internist to women taking potentially teratogenic medications. Many internists in the Eisenberg study believed that an EMR alert would be worthwhile. In addition, approximately two-thirds of the internists in the Eisenberg study agreed that "a referral or telephone consultation service for assistance in providing appropriate contraception for women on potential teratogens would be useful." In order to improve the contraceptive counseling among women prescribed potentially teratogenic medications, the investigators for the proposed project have been conducting collaborative research for the past two years with the Family Medicine and the California Teratogen Information Service (CTIS). First, the investigators conducted a cross-sectional study to assess contraceptive utilization among women prescribed category D or X medications. Investigators obtained access to the EMR of women seen in an academic Family Medicine Department between April 2011 to April 2012 who were taking a category D or X medication. Information was abstracted regarding the specific category D or X medication, demographics, sexual activity and the contraceptive method. There were a total of 610 women included in this study. Among the 610 women, 72 (11.8%) of women had documentation in the EMR that they were not asked about their sexual activity. Sexual activity with men was documented in 407 of the 610 women. Of the 407 women who were sexually active with men, 132 (32.4%) had no contraceptive method documented in the EMR. Despite the importance of avoiding an unintended pregnancy in women taking teratogens, the contraceptive utilization rate is similar to the national average (38% of 15-44 year olds reported not using a contraceptive method). In addition, among the women using contraception, the most common contraceptive method was oral contraceptives, which is very user dependent with a typical failure rate of 9%. In fact, the oral contraceptive compliance rate for women taking teratogens is the same as the national compliance rate.

Next, we conducted a descriptive pilot study to evaluate the feasibility and patient satisfaction with an EMR alert and referral system. This intervention was chosen since the Eisenberg study identified the time constraint issue, the acceptability of EMR alert, and the acceptability of the telephone consultation service. Women of reproductive age who were seen by a Family Medicine clinician at a UCSD Medical Center clinic with access to the EMR were included in the pilot study. If a woman of reproductive age was seen by a Family Medicine clinician and she was currently taking or was newly prescribed a category D or X medications, an EMR electronic alert was be generated for the clinician. The alert said "This patient may benefit from a referral to the CTIS Information Line for counseling," click "Accept" or "Decline". The alert was purposefully created so it is easier to accept the referral. If the Family Medicine clinician clicked "Decline" then a reason must be given for declining the referral. If the clinician decided a referral is appropriate, he/she clicked "Accept" and informed the patient that she will be contacted by CTIS. The referral was also included in the patient instructions.

Within one month of the referral, a CTIS counselor contacted the patient and reviewed the category D or X medication and potential effects if the patient were to become pregnant as well as contraceptive options. The counseling included some information about the efficacy of each contraceptive method. She was instructed that she could return to her Family Medicine clinician for contraceptive service delivery. She was also offered a referral to Reproductive Medicine at UCSD for further counseling. The referring Family Medicine clinician was then informed of the outcome of the referral via an EMR communication. Following counseling a phone interview was used to assess contraceptive utilization and motivation. In addition a satisfaction survey completed. Contraceptive utilization was assessed using a modified version of Module 5 of Behavioral Risk Factor Surveillance System. Participant satisfaction was assessed using a Likert scale.

Among 25 participants in the pilot study, 11 (44%) women were using oral contraceptives, 7 (28%) women were using condoms, 3 (12%) women were using withdrawal, 2 (8%) women were using the IUD, 1 (4%) woman was using vaginal contraceptive ring and 1 (4%) woman was not using contraception. Among the women using oral contraceptive, the majority of the women underestimated the typical failure rate. Among the women using contraception, only 2 women stated that they chose their current contraceptive method based on the effectiveness in preventing pregnancy. After receiving the teratogen and contraceptive counseling, 25% of women using contraception were considering using a more effective contraceptive method. The women were also asked about when they would want a child, the most common response was wanting a child in 2-5 years. Satisfaction with the referral system and counseling was high. Approximately 96% of participants strongly agreed or agreed that the information they received on contraceptive options was helpful.

The conclusion from this descriptive pilot study is that an EMR referral system for teratogen and contraceptive counseling for women prescribed category D or X medications is feasible and has high patient satisfaction. Women taking category D or X medications are not currently choosing a contraceptive method based on efficacy of preventing pregnancy, therefore efficacy should emphasized more in future contraceptive counseling interventions. Most participants indicated that they wanted a child in 2-5 years. The results of this pilot study support promoting long-acting reversible contraception in this population. In addition, the pilot study revealed that the contraceptive counseling can motivate women taking potentially teratogenic medications to consider using more effective contraception. Now we need to focus on helping these women go from thinking about using more effective to actually using more effective contraception.

The proposed project incorporates the findings of this pilot study to facilitate intention to use more effective contraception into behavior change. It utilizes the EMR to not only identify and counsel women exposed to high risk medications, but also facilitates behavior change by incorporating a clinic visit to further discuss and receive more effective contraception. The primary objective for the study is to determine if an EMR referral to teratogen counseling, contraceptive counseling and a follow up contraceptive appointment will increase the utilization of more effective contraception among women prescribed category D or X medications. The Internal Medicine department and Family Medicine department have approved the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Background: No limitation, will include minorities and Spanish speaking participants
* Health Status: no limitation
* Sexually active with men
* Currently taking the Category D or X medication

Exclusion Criteria:

* Currently Pregnant
* Not currently sexually active with men
* History of hysterectomy, bilateral oophorectomy, history of female sterilization
* Partner with history of vasectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Utilization of More Effective Contraception | 1 year
  Change of contraception from baseline questionnaire compared to 3 and 6 month follow up with improved contraception defined as 1) no contraception changed to some form of contraception, 2) barrier methods changed to combined hormonal contraception/ IUD/contraceptive implant/tubal ligation, or 3) combined hormonal method to an IUD/contraceptive implant/tubal ligation.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD MPH, Principal Investigator — UCSD Department of Reproductive Medicine
Locations (1):
- CTIS Pregnancy Health Information Line at the University of California San Diego, San Diego, California, United States

REFERENCES:
- [Background] Santucci AK, Gold MA, Akers AY, Borrero S, Schwarz EB. Women's perspectives on counseling about risks for medication-induced birth defects. Birth Defects Res A Clin Mol Teratol. 2010 Jan;88(1):64-9. doi: 10.1002/bdra.20618. PMID 19637252
- [Background] Eisenberg DL, Stika C, Desai A, Baker D, Yost KJ. Providing contraception for women taking potentially teratogenic medications: a survey of internal medicine physicians' knowledge, attitudes and barriers. J Gen Intern Med. 2010 Apr;25(4):291-7. doi: 10.1007/s11606-009-1215-2. Epub 2010 Jan 20. PMID 20087677
- [Background] Jones J, Mosher W, Daniels K. Current contraceptive use in the United States, 2006-2010, and changes in patterns of use since 1995. Natl Health Stat Report. 2012 Oct 18;(60):1-25. PMID 24988814
- [Background] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Background] Steinkellner A, Chen W, Denison SE. Adherence to oral contraception in women on Category X medications. Am J Med. 2010 Oct;123(10):929-934.e1. doi: 10.1016/j.amjmed.2010.05.009. PMID 20920695